CLINICAL TRIAL: NCT03064126
Title: RANGER II SFA: A 3:1 Randomized Trial Comparing the Boston Scientific RANGER™ Paclitaxel Coated Balloon vs Standard Balloon Angioplasty for the Treatment of Superficial Femoral Arteries (SFA) and Proximal Popliteal Arteries (PPA)
Brief Title: RANGER™ Paclitaxel Coated Balloon vs Standard Balloon Angioplasty
Acronym: RANGER II SFA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2062
Record Dates: First submitted 2017-01-13; First posted 2017-02-24 (Actual); Results first posted 2020-07-15 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Artery Disease; Atherosclerosis; Artery Diseases, Peripheral; Plaque, Atherosclerotic; Occlusive Arterial Disease
Keywords: Artery; Atherosclerosis; Arterial; Peripheral; Plaque; Angioplasty; PTA
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis; Plaque, Atherosclerotic; Arterial Occlusive Diseases; Plaque, Amyloid | interventions — Angioplasty; Paclitaxel

STUDY DESIGN:
Intervention Model Description: The RANGER™ investigational device is coated with the drug paclitaxel.
Who Masked: Participant
Masking Description: Subjects will be blinded to treatment assigned and treatment received until completion of all 12 month follow-up visits (primary endpoint).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- RANGER™ Paclitaxel Coated Balloon (Experimental): RANGER™ Paclitaxel Coated Balloon Catheter angioplasty in the SFA/PPA at the index procedure.
  Subjects will be randomized 3:1 to the drug coated or standard angioplasty balloon.
  Interventions: Device: RANGER™ Paclitaxel Coated Balloon; Drug: Paclitaxel
- Standard Balloon Angioplasty (Active Comparator): Standard Balloon Catheter angioplasty in the SFA/PPA at the index procedure. Subjects will be randomized 3:1 to the drug coated or standard angioplasty balloon.
  Interventions: Procedure: Standard Balloon Angioplasty

INTERVENTIONS:
Device: RANGER™ Paclitaxel Coated Balloon — A procedure that utilizes a balloon coated with paclitaxel (drug) which can open up a blocked blood vessel using a small, flexible plastic tube, or catheter, with a "balloon" at the end of it. When the tube is in place, it inflates to open the blood vessel, or artery, so that normal blood flow is restored. The tube is then removed. The blood vessels that will be treated in the RANGER II SFA study include the superficial femoral arteries and the proximal popliteal arteries.
  Other Names: Percutaneous Transluminal Angioplasty (PTA)
  Arms: RANGER™ Paclitaxel Coated Balloon
Drug: Paclitaxel — The RANGER™ Balloon is coated with the drug Paclitaxel.
  Arms: RANGER™ Paclitaxel Coated Balloon
Procedure: Standard Balloon Angioplasty — A procedure that utilizes an uncoated balloon which can open up a blocked blood vessel using a small, flexible plastic tube, or catheter, with a "balloon" at the end of it. When the tube is in place, it inflates to open the blood vessel, or artery, so that normal blood flow is restored. The tube is then removed. The blood vessels that will be treated in the RANGER II SFA study include the superficial femoral arteries and the proximal popliteal arteries.
  Other Names: Percutaneous Transluminal Angioplasty (PTA)
  Arms: Standard Balloon Angioplasty

SUMMARY:
To evaluate the safety and effectiveness of the Ranger™ Paclitaxel Coated Balloon for treating lesions located in the superficial femoral and proximal popliteal arteries (SFA/PPA).

Long Balloon substudy: To evaluate the safety and effectiveness of the Boston Scientific Corporation (BSC) Ranger™ Paclitaxel Coated Balloon in the 120, 150 and 200 mm lengths for treating Superficial Femoral Artery (SFA) and/or Proximal Popliteal Artery (PPA) lesions.

DETAILED DESCRIPTION:
The RANGER II SFA is a global, prospective, multi-center clinical trial. Approximately 446 subjects will be enrolled at up to 80 study centers worldwide. Regions participating include the United States, Canada, European Union, Japan and New Zealand.

The trial consists of a single-blind, superiority, 3:1 (Ranger Drug-Coated Balloon (DCB) vs. Standard PTA) randomized controlled trial (RCT) and a concurrent, non-randomized, single-arm, pharmacokinetic (PK) substudy, and a concurrent, non-blinded, non-randomized, Long balloon substudy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject (or Legal Guardian) is willing and able to provide consent before any study-specific tests or procedures are performed and agree to attend all required follow-up visits;
2. Subject at least 20 years of age;
3. Chronic symptomatic lower limb ischemia defined as Rutherford classification 2, 3, or 4;
4. Target lesion is in the native SFA and/or PPA down to the P1 segment;
5. Patent popliteal and infrapopliteal arteries, i.e., single vessel runoff or better with at least one of three vessels patent (less than 50 % stenosis) to the ankle or foot;
6. Reference vessel diameter ≥ 4 mm and ≤ 8 mm by visual estimate;
7. Angiographic evidence that target lesion consists of a single de novo, non-stented and non-atherectomy treated or restenotic lesion (or tandem lesions or a combination lesion as defined below) that is:

   * ≥ 70%-99% stenotic with total lesion length up to 180 mm by visual estimate.
   * Occluded with total lesion length ≤ 100 mm by visual estimate.
   * If lesion is restenotic, most recent PTA treatment must be > 3 months prior to enrollment.

Exclusion Criteria:

1. Life expectancy, documented in the Investigator's opinion, of less than 12 months;
2. Hemorrhagic stroke or cardiac event (e.g. STEMI, unstable angina) within 6 months prior to enrollment;
3. Known allergies or sensitivities to heparin, aspirin, other anticoagulant/antiplatelet therapies, and/or paclitaxel;
4. Known hypersensitivity or contraindication to contrast dye that, in the opinion of the investigator, cannot be adequately pre-medicated;
5. Chronic renal insufficiency with serum creatinine > 2.0 mg/dL within 30 days of index procedure or treatment with dialysis;
6. Platelet count < 80,000 mm 3 or > 600,000 mm 3 or history of bleeding diathesis;
7. Receiving immunosuppressive therapy;
8. Septicemia at the time of enrollment;
9. Any major intervention planned within 30 days post index procedure;
10. Presence of other hemodynamically significant outflow lesions in the target limb requiring intervention within 30 days of enrollment;
11. Failure to successfully cross the target lesion with a guidewire;
12. Failure to successfully pre-dilate the target vessel;
13. Patient has lesion that requires the use of adjunctive primary treatment modalities (i.e. laser, atherectomy, scoring/cutting balloon, other debulking devices, etc.) during the index procedure;
14. History of major amputation in the target limb;
15. Target lesion or vessel has ever been previously treated with stent (e.g. in-stent restenosis) or surgery. Target lesion or vessel has been treated with atherectomy or a DCB in the past 12 months;
16. Pregnant or breast feeding;
17. Presence of aneurysm in the target vessel;
18. Acute ischemia and/or acute thrombosis of the SFA/PPA prior to enrollment;
19. Patient has significant inflow disease which cannot be treated prior to the target lesion treatment;
20. Patient has perforated targeted vessel as evidenced by extravasation of contrast media;
21. Patient has severe calcification that renders the lesion undilatable;
22. Current participation in another investigational drug or device clinical trial that has not completed the primary endpoint at the time of randomization/enrollment or that clinically interferes with the current trial endpoints.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2023-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, MD, Principal Investigator — Universitaets-Herzzentrum; Ravish Sachar, MD, Principal Investigator — University of North Carolina - Rex Hospital
Locations (67):
- United States (42):
  - Thomas Hospital, Fairhope, Alabama
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - The Vascular Experts, Stratford, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - South Florida Vascular Associates, Coconut Creek, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth Sebring, Sebring, Florida
  - Wellstar Hospitals, Marietta, Georgia
  - Kaiser Foundation Hospitals, Honolulu, Hawaii
  - St. Joseph Hospital, Fort Wayne, Indiana
  - Community Hospital, Munster, Indiana
  - King's Daughters Medical Center - Kentucky Heart Institute, Ashland, Kentucky
  - Terrebonne General Medical Center, Houma, Louisiana
  - Mercy Hospital, Coon Rapids, Minnesota
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - Rex Hospital, Raleigh, North Carolina
  - Coastal Carolina Surgical Associates, Wilmington, North Carolina
  - Bethesda North Hospital, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Premier Cardiovascular Institute, Dayton, Ohio
  - Northeast Ohio Vascular Associates, Inc., Willoughby, Ohio
  - St. Charles Medical Center, Bend, Oregon
  - Temple University, Philadelphia, Pennsylvania
  - University Medical Center-Greenville Memorial Hospital, Greenville, South Carolina
  - Turkey Creek Medical Center, Knoxville, Tennessee
  - North Park Heart & Vascular Center, Dallas, Texas
  - Cardiology Clinic of San Antonio, Live Oak, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - North Dallas Research Associates, McKinney, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - THR Presbyterian Plano, Plano, Texas
  - Tyler Cardiac and Endovascular Center, Tyler, Texas
  - Davis Hospital and Medical Center, Layton, Utah
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Aspirus Heart and Vascular Institute, Wausau, Wisconsin
- Austria (3):
  - Medizinische Univ.-Kliniken Graz, Graz
  - Allgemeines Krankenhaus AKH, Vienna
  - Hanusch-Krankenhaus, Vienna
- Belgium (3):
  - Ziekenhuis Oost Limburg, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - Regionaal Ziekenhuis Heilig Hart Tienen, Tienen
- Canada (4):
  - Peter Lougheed Centre, Calgary, Alberta
  - Hamilton General Hospital, Hamilton, Ontario
  - Fleurimont Hospital, Sherbrooke, Quebec
  - Hopital Saint - Francois d'Assise, Québec
- Japan (12):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Iwaki City Medical Center, Iwaki, Fukushima
  - Tokeidai Memorial Hospital, Sapporo, Hokkaido
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Saiseikai Yokohama-City Eastern Hospital, Yokohama, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Kasukabe Chuo General Hospital, Kasukabe, Saitama
  - Saiseikai Central Hospital, Minato, Tokyo
  - Kyoto Katsura Hospital, Kyoto
  - Morinomiya Hospital, Osaka
  - Osaka Saiseikai Nakatsu Hospital, Osaka
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Clinical Trials NZ, Hamilton
  - Middlemore Hospital, Otahuhu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Litsky J, Chanda A, Stilp E, Lansky A, Mena C. Critical evaluation of stents in the peripheral arterial disease of the superficial femoral artery - focus on the paclitaxel eluting stent. Med Devices (Auckl). 2014 May 28;7:149-56. doi: 10.2147/MDER.S45472. eCollection 2014. PMID 24920940
- [Background] Kakkar AM, Abbott JD. Percutaneous versus surgical management of lower extremity peripheral artery disease. Curr Atheroscler Rep. 2015;17(2):479. doi: 10.1007/s11883-014-0479-0. PMID 25612856
- [Background] Razavi MK, Mustapha JA, Miller LE. Contemporary systematic review and meta-analysis of early outcomes with percutaneous treatment for infrapopliteal atherosclerotic disease. J Vasc Interv Radiol. 2014 Oct;25(10):1489-96, 1496.e1-3. doi: 10.1016/j.jvir.2014.06.018. Epub 2014 Aug 15. PMID 25130307
- [Background] Laird JR, Katzen BT, Scheinert D, Lammer J, Carpenter J, Buchbinder M, Dave R, Ansel G, Lansky A, Cristea E, Collins TJ, Goldstein J, Jaff MR; RESILIENT Investigators. Nitinol stent implantation versus balloon angioplasty for lesions in the superficial femoral artery and proximal popliteal artery: twelve-month results from the RESILIENT randomized trial. Circ Cardiovasc Interv. 2010 Jun 1;3(3):267-76. doi: 10.1161/CIRCINTERVENTIONS.109.903468. Epub 2010 May 18. PMID 20484101
- [Background] Scheinert D, Duda S, Zeller T, Krankenberg H, Ricke J, Bosiers M, Tepe G, Naisbitt S, Rosenfield K. The LEVANT I (Lutonix paclitaxel-coated balloon for the prevention of femoropopliteal restenosis) trial for femoropopliteal revascularization: first-in-human randomized trial of low-dose drug-coated balloon versus uncoated balloon angioplasty. JACC Cardiovasc Interv. 2014 Jan;7(1):10-9. doi: 10.1016/j.jcin.2013.05.022. PMID 24456716
- [Derived] Schroe H, Sachar R, Keirse K, Soga Y, Brodmann M, Rao V, Werner M, Holden A, Lopez L, Krishnan P, Diaz-Cartelle J. The RANGER II superficial femoral artery trial: 1-year results of the long lesion cohort. Vasc Med. 2022 Oct;27(5):457-465. doi: 10.1177/1358863X221097164. Epub 2022 Aug 9. PMID 35943120
- [Derived] Soga Y, Fujihara M, Yamamoto Y, Nakamura S, Iida O, Kawasaki D, Urasawa K, Ando H, Mori S, Suzuki K, Horie K, Diaz-Cartelle J, Kozuki A. One-year results for Japanese patients in RANGER II SFA. Heart Vessels. 2022 Apr;37(4):568-573. doi: 10.1007/s00380-021-01947-3. Epub 2021 Sep 23. PMID 34557931
- [Derived] Sachar R, Soga Y, Ansari MM, Kozuki A, Lopez L, Brodmann M, Schroe H, Ramanath VS, Diaz-Cartelle J, Zeller T; RANGER II SFA Investigators. 1-Year Results From the RANGER II SFA Randomized Trial of the Ranger Drug-Coated Balloon. JACC Cardiovasc Interv. 2021 May 24;14(10):1123-1133. doi: 10.1016/j.jcin.2021.03.021. PMID 34016410

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 440 subjects were enrolled in the trial (376 subjects in the Randomized Controlled Trial (RCT), 52 subjects in the Long Balloon (LB) substudy and 12 subjects in the Pharmacokinetic (PK) substudy). RCT subjects were randomized to Ranger Drug-Coated Balloon (DCB) or Standard Percutaneous Transluminal Angioplasty (PTA) at a 3:1 ratio, respectively. All LB and PK subjects were treated with the Ranger DCB. RCT/PK shows 60 months data; LB shows 12 month data.
Groups:
- RANGER™ Paclitaxel Coated Balloon RCT: RANGER™ Paclitaxel Coated Balloon Catheter angioplasty in the SFA/PPA at the index procedure.
  Subjects will be randomized 3:1 to the drug coated or standard angioplasty balloon.
  RANGER™ Paclitaxel Coated Balloon: A procedure that utilizes a balloon coated with paclitaxel (drug) which can open up a blocked blood vessel using a small, flexible plastic tube, or catheter, with a "balloon" at the end of it. When the tube is in place, it inflates to open the blood vessel, or artery, so that normal blood flow is restored. The tube is then removed. The blood vessels that will be treated in the RANGER II SFA study include the superficial femoral arteries and the proximal popliteal arteries.
  Paclitaxel: The RANGER™ Balloon is coated with the drug Paclitaxel.
- Standard Balloon Angioplasty RCT: Standard Balloon Catheter angioplasty in the SFA/PPA at the index procedure. Subjects will be randomized 3:1 to the drug coated or standard angioplasty balloon.
  Standard Balloon Angioplasty: A procedure that utilizes an uncoated balloon which can open up a blocked blood vessel using a small, flexible plastic tube, or catheter, with a "balloon" at the end of it. When the tube is in place, it inflates to open the blood vessel, or artery, so that normal blood flow is restored. The tube is then removed. The blood vessels that will be treated in the RANGER II SFA study include the superficial femoral arteries and the proximal popliteal arteries.
- Long Balloon (LB) Substudy: The Long Balloon substudy cohort will evaluate the safety and effectiveness of the Ranger DCB in the 120, 150 and 200 mm lengths for treating SFA and/or PPA lesions.
- Pharmacokinetics (PK) Substudy: The PK substudy cohort will evaluate the safety and pharmacokinetics of the levels of paclitaxel in the systemic circulation of subjects at multiple time points after treatment with the Ranger DCB. Time points for analysis are a venous blood draw at screening, followed by blood draws at 10 minutes, 30 minutes, 1 hour, 3 hours, 6 hours and 24 or 48 hours after last Ranger DCB balloon removal, as well as 7 days and 30 days post index procedure.
Period: Overall Study
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT | Long Balloon (LB) Substudy | Pharmacokinetics (PK) Substudy
Started | 278 | 98 | 52 | 12
Completed | 203 | 67 | 48 | 8
Not Completed | 75 | 31 | 4 | 4
Not completed — Death | 40 | 16 | 4 | 2
Not completed — Withdrawal by Subject | 17 | 9 | 0 | 2
Not completed — Lost to Follow-up | 7 | 3 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 0 | 0
Not completed — Other reason for early termination | 3 | 2 | 0 | 0
Not completed — Missed Visit | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- RANGER™ Paclitaxel Coated Balloon RCT: RANGER™ Paclitaxel Coated Balloon Catheter angioplasty in the SFA/PPA at the index procedure.
- Standard Balloon Angioplasty RCT: Standard Balloon Catheter angioplasty in the SFA/PPA at the index procedure.
- Total: Total of all reporting groups
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT | Long Balloon (LB) Substudy | Pharmacokinetics (PK) Substudy | Total
Number analyzed (Participants) | 278 | 98 | 52 | 12 | 440
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.6 (9.5) | 69.1 (10.3) | 70.3 (9.9) | 63.3 (13.3) | 70.06 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 31 | 14 | 8 | 158
  Male | 173 | 67 | 38 | 4 | 282
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 8 | 0 | 0 | 29
  Caucasian | 155 | 59 | 51 | 9 | 274
  Asian (Japanese) | 77 | 25 | 0 | 0 | 102
  Black, or African Heritage | 20 | 4 | 1 | 3 | 28
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Other | 1 | 0 | 0 | 0 | 1
  Not Disclosed | 3 | 2 | 0 | 0 | 5
Region of Enrollment [Number; unit: participants]
  New Zealand | 7 | 2 | 2 | 0 | 11
  Canada | 12 | 4 | 0 | 0 | 16
  Europe | 29 | 8 | 50 | 0 | 87
  Japan | 77 | 25 | 0 | 0 | 102
  United States | 153 | 59 | 0 | 12 | 224
History of Smoking (Current) [Count of Participants; unit: Participants] | 87 | 45 | 24 | 6 | 162
History of Smoking (Previous) [Count of Participants; unit: Participants] | 150 | 38 | 23 | 5 | 216
History of Smoking (Never) [Count of Participants; unit: Participants] | 40 | 15 | 5 | 1 | 61
History of Smoking (Unknown) [Count of Participants; unit: Participants] | 1 | 0 | 0 | 0 | 1
Current Diabetes Mellitus [Count of Participants; unit: Participants] | 118 | 43 | 17 | 8 | 186
History of Hyperlipidemia requiring medication [Count of Participants; unit: Participants] — Population: History of Hyperlipidemia requiring medication rates are based on number of evaluable subjects - subjects with the data point collected.
  Participants
    number analyzed (Participants) | 278 | 98 | 51 | 12 | 439
    (all) | 211 | 78 | 42 | 10 | 341
History of Hypertension requiring medication [Count of Participants; unit: Participants] | 251 | 80 | 37 | 9 | 377
History of Chronic Obstructive Pulmonary Disease [Count of Participants; unit: Participants] — Population: History of Chronic Obstructive Pulmonary Disease rates are based on number of evaluable subjects - subjects with the data point collected.
  Participants
    number analyzed (Participants) | 275 | 98 | 50 | 12 | 435
    (all) | 52 | 21 | 9 | 2 | 84
History of Coronary Artery Disease (CAD) [Count of Participants; unit: Participants] — Population: History of Coronary Artery Disease rates are based on number of evaluable subjects - subjects with the data point collected.
  Participants
    number analyzed (Participants) | 276 | 98 | 52 | 12 | 438
    (all) | 131 | 44 | 14 | 7 | 196
History of Myocardial Infarction (MI) [Count of Participants; unit: Participants] — Population: History of Myocardial Infarction rates are based on number of evaluable subjects - subjects with the data point collected.
  Participants
    number analyzed (Participants) | 277 | 97 | 52 | 12 | 438
    (all) | 46 | 14 | 6 | 4 | 70
History of Congestive Heart Failure (CHF) [Count of Participants; unit: Participants] — Population: History of Congestive Heart Failure rates are based on number of evaluable subjects - subjects with the data point collected.
  Participants
    number analyzed (Participants) | 277 | 98 | 51 | 12 | 438
    (all) | 26 | 9 | 1 | 0 | 36
NYHA Classification [Count of Participants; unit: Participants] — Population: NYHA classification rates are based on number of evaluable subjects - subjects with the data point collected.
  Participants
    number analyzed (Participants) | 26 | 9 | 1 | 0 | 36
    NYHA I Classification | 10 | 0 | 0 |  | 10
    NYHA II Classification | 6 | 6 | 0 |  | 12
    NYHA III Classification | 1 | 0 | 0 |  | 1
    NYHA IV Classification | 0 | 0 | 0 |  | 0
    NYHA Unknown Classification | 9 | 3 | 1 |  | 13
History of Percutaneous Coronary Intervention (PCI) [Count of Participants; unit: Participants] — Population: History of Percutaneous Coronary Intervention rates are based on number of evaluable subjects - subjects with the data point collected.
  Participants
    number analyzed (Participants) | 274 | 98 | 51 | 12 | 435
    (all) | 81 | 34 | 8 | 2 | 125
History of Coronary Artery Bypass Graft (CABG) Surgery [Count of Participants; unit: Participants] — Population: History of Coronary Artery Bypass Graft rates are based on number of evaluable subjects - subjects with the data point collected.
  Participants
    number analyzed (Participants) | 277 | 97 | 52 | 12 | 438
    (all) | 35 | 15 | 1 | 1 | 52
Stable Angina [Count of Participants; unit: Participants] | 35 | 13 | 1 | 0 | 49
Unstable Angina [Count of Participants; unit: Participants] | 1 | 0 | 0 | 0 | 1
No Angina [Count of Participants; unit: Participants] | 242 | 85 | 50 | 12 | 389
Angina (Unknown) [Count of Participants; unit: Participants] | 0 | 0 | 1 | 0 | 1
History of Transient Ischemic Attacks (TIA) [Count of Participants; unit: Participants] — Population: History of Transient Ischemic Attacks rates are based on number of evaluable subjects - subjects with the data point collected.
  Participants
    number analyzed (Participants) | 275 | 97 | 52 | 12 | 436
    (all) | 14 | 7 | 5 | 0 | 26
History of Cerebrovascular Accident (CVA) [Count of Participants; unit: Participants] — Population: History of Cerebrovascular Accident rates are based on number of evaluable subjects - subjects with the data point collected.
  Participants
    number analyzed (Participants) | 276 | 98 | 52 | 12 | 438
    (all) | 36 | 11 | 2 | 2 | 51
History of Renal Insufficiency [Count of Participants; unit: Participants] — Population: History of Renal Insufficiency rates are based on number of evaluable subjects - subjects with the data point collected.
  Participants
    number analyzed (Participants) | 278 | 97 | 52 | 12 | 439
    (all) | 30 | 5 | 6 | 3 | 44
History of Renal Percutaneous Intervention [Count of Participants; unit: Participants] — Population: History of Renal Percutaneous Intervention rates are based on number of evaluable subjects - subjects with the data point collected.
  Participants
    number analyzed (Participants) | 275 | 97 | 52 | 12 | 436
    (all) | 6 | 1 | 0 | 0 | 7
History of Peripheral Vascular Surgery [Count of Participants; unit: Participants] — Population: History of Peripheral Vascular Surgery rates are based on number of evaluable subjects - subjects with the data point collected.
  Participants
    number analyzed (Participants) | 277 | 98 | 52 | 12 | 439
    (all) | 24 | 9 | 8 | 0 | 41
History of Endovascular Interventions [Count of Participants; unit: Participants] — Population: History of Endovascular Interventions rates are based on number of evaluable subjects - subjects with the data point collected.
  Participants
    number analyzed (Participants) | 278 | 97 | 52 | 12 | 439
    (all) | 131 | 47 | 23 | 4 | 205
History of Claudication [Count of Participants; unit: Participants] | 271 | 90 | 50 | 12 | 423

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Primary Lesion Patency
Description: RCT outcome measure: Primary patency of the target lesion is determined by Peak Systolic Velocity Ratio (PSVR) ≤ 2.4 (by duplex ultrasound (DUS)) and freedom from clinically-driven Target Lesion Revascularization (TLR) within 12 months from procedure. Lesion patency is defined as freedom from more than 50% stenosis based on DUS PSVR comparing data within the treated segment to the proximal normal arterial segment. PSVR >2.4 suggests >50% stenosis.
  LB Substudy outcome measure: Primary patency of the target lesion is determined by duplex ultrasound (DUS) peak systolic velocity ratio (PSVR) ≤ 2.4 in absence of clinically-driven TLR. Primary effectiveness endpoint is assessed at 6 months post-procedure.
  PK Substudy: There was no prespecified analysis of primary lesion patency.
Time Frame: 12 months (RCT); 6 months (LB substudy)
Population: Percentage (%) of lesions that reach endpoint without a hemodynamically significant stenosis on DUS and without clinically-driven TLR or bypass of the target lesion.
  PK Substudy: There was no prespecified analysis of primary lesion patency.
Measure: Count of Participants; unit: Participants
Groups:
- Long Balloon (LB) Substudy: The Long Balloon substudy cohort will evaluate the safety and effectiveness of the Ranger DCB in the 120, 150 and 200 mm lengths for treating SFA and/or PPA lesions.
  Primary safety and effectiveness endpoints for the LB Substudy are assessed at 6 months post-procedure.
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT | Long Balloon (LB) Substudy
Number analyzed (Participants) | 234 | 86 | 46
Participants | 194 | 57 | 43
Statistical Analysis 1: Comparison: RANGER™ Paclitaxel Coated Balloon RCT vs Standard Balloon Angioplasty RCT; Test type: Superiority; p = 0.0017, Chi-squared; Risk Difference (RD) = 0.166, 97.5% CI 1-sided [lower limit 0.0553]

2. Primary Outcome: Major Adverse Events (MAEs) (Primary Safety Endpoint)
Description: RCT: MAE is defined as a composite of freedom from all-cause death through 1 month, target limb major amputation (defined as at or above the ankle) within 12 months, and/or Target Lesion Revascularization (TLR) within 12 months.
  LB Substudy: Primary safety endpoint assesses the occurrence of MAE defined as all-cause death through 1 month, target limb major amputation and/or TLR at 6 and 12 months post-index procedure.
  PK Substudy: There was no prespecified analysis of primary safety endpoint.
Time Frame: Primary safety endpoint assessed at 12 months for RCT study and at both 6 and 12 months for LB substudy.
Population: PK Substudy: There was no prespecified analysis of primary safety endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT | Long Balloon (LB) Substudy
Number analyzed (Participants) | 278 | 98 | 52
Participants
  6 Month Primary Safety Endpoint: number analyzed (Participants) | 0 | 0 | 52
  6 Month Primary Safety Endpoint |  |  | 50
  12 Month Primary Safety Endpoint: number analyzed (Participants) | 256 | 91 | 50
  12 Month Primary Safety Endpoint | 241 | 76 | 47
Statistical Analysis 1: Comparison: RANGER™ Paclitaxel Coated Balloon RCT vs Standard Balloon Angioplasty RCT; Test type: Non-Inferiority — A Chi-Square Test was used to assess the hypothesis for the difference in 12-month MAE-free rate with non-inferiority margin (-10%); p < 0.0001, Chi-squared; Risk Difference (RD) = 0.106, 97.5% CI 1-sided [lower limit 0.0248]

3. Secondary Outcome: Number of Participants With Technical Success of Angioplasty Procedure
Description: Technical success defined as successful delivery, balloon inflation and deflation and retrieval of the intact trial device without burst below the rated burst pressure.
  RCT Standard Balloon Angioplasty: Device deficiency data is only collected for Ranger DCB; data not collected for Standard PTA group; there is no pre-specified analysis of this outcome for the Standard PTA group.
Time Frame: Day 0
Population: RCT: Device deficiency data is only collected for Ranger DCB; data not collected for Standard PTA group; there is no pre-specified analysis of this outcome for the Standard PTA group.
Measure: Count of Participants; unit: Participants
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT | Long Balloon (LB) Substudy | Pharmacokinetics (PK) Substudy
Number analyzed (Participants) | 278 | 0 | 52 | 12
Participants | 277 |  | 47 | 12

4. Secondary Outcome: Number of Participants With Procedural Success of Angioplasty Procedure
Description: Procedural success defined as residual stenosis of less than or equal to 50% (non-stented subjects) or less than or equal to 30% (stented subjects) by core laboratory evaluation.
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT | Long Balloon (LB) Substudy | Pharmacokinetics (PK) Substudy
Number analyzed (Participants) | 278 | 98 | 52 | 12
Participants | 269 | 97 | 49 | 12

5. Secondary Outcome: Number of Participants With Clinical Success Rate Assessment
Description: Clinical success defined as procedural success without procedural complications including death, major target limb amputation, thrombosis of the target lesion, or clinically-driven TLR prior to discharge.
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT | Long Balloon (LB) Substudy | Pharmacokinetics (PK) Substudy
Number analyzed (Participants) | 278 | 98 | 52 | 12
Participants | 267 | 96 | 48 | 11

6. Secondary Outcome: Number of Major Adverse Event (MAE) Assessment
Description: MAEs defined as all-cause of death post-index procedure (30-days), target limb major amputation, and/or target lesion revascularization (TLR) through 60-months in RCT.
  MAEs defined as all-cause of death post-index procedure (30-days), target limb major amputation, and/or target lesion revascularization (TLR) through 12-months in LB substudy.
  PK Substudy: There was no prespecified analysis of MAEs for PK substudy.
Time Frame: 60-months (RCT); 12-months (LB substudy).
Population: MAE assessment rates are based on number of evaluable subjects - subjects with the data point collected.
  PK Substudy: There was no prespecified analysis of MAEs for PK substudy.
Measure: Count of Participants; unit: Participants
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT | Long Balloon (LB) Substudy
Number analyzed (Participants) | 278 | 98 | 52
Participants
  12-Month MAE (Composite Endpoint): number analyzed (Participants) | 256 | 91 | 50
  12-Month MAE (Composite Endpoint) | 15 | 15 | 3
  12-Month All Causes of Death at 1-Month: number analyzed (Participants) | 256 | 91 | 50
  12-Month All Causes of Death at 1-Month | 1 | 0 | 0
  12-Month Target Limb Major Amputation: number analyzed (Participants) | 256 | 91 | 50
  12-Month Target Limb Major Amputation | 0 | 0 | 0
  12-Month Target Lesion Revascularization: number analyzed (Participants) | 256 | 91 | 50
  12-Month Target Lesion Revascularization | 14 | 15 | 3
  60-Month MAE (Composite Endpoint): number analyzed (Participants) | 213 | 73 | 0
  60-Month MAE (Composite Endpoint) | 57 | 23 |
  60-Month All Causes of Death at 1-Month: number analyzed (Participants) | 213 | 73 | 0
  60-Month All Causes of Death at 1-Month | 1 | 0 |
  60-Month Target Limb Major Amputation: number analyzed (Participants) | 213 | 73 | 0
  60-Month Target Limb Major Amputation | 1 | 0 |
  60-Month Target Lesion Revascularization: number analyzed (Participants) | 213 | 73 | 0
  60-Month Target Lesion Revascularization | 56 | 23 |

7. Secondary Outcome: Number of Clinical Events Committee (CEC) Adjudicated Events
Description: CEC adjudicated events including death of any cause, target lesion revascularization (TLR), target vessel revascularization (TVR) and target limb amputation (TLA).
  Denominators for the cumulative rate will be based on 1) subjects with events, and 2) subjects with no events but their follow-up time reaches (or is beyond) the earliest visit window.
  LB substudy follow-up through 12 month.
Time Frame: 1, 6, 12, 24, 36, 48 and 60 months (RCT and PK substudy); 1, 6 and 12 months (LB substudy)
Population: Denominators for the cumulative rate will be based on 1) subjects with events, and 2) subjects with no events but their follow-up time reaches (or is beyond) the earliest visit window.
Measure: Number; unit: Participants
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT | Long Balloon (LB) Substudy | Pharmacokinetics (PK) Substudy
Number analyzed (Participants) | 278 | 98 | 52 | 12
Participants
  1-Month All Deaths: number analyzed (Participants) | 277 | 98 | 52 | 12
  1-Month All Deaths | 1 | 0 | 0 | 0
  1-Month All Target Lesion Revascularization (TLR): number analyzed (Participants) | 277 | 98 | 52 | 12
  1-Month All Target Lesion Revascularization (TLR) | 0 | 0 | 1 | 0
  1-Month All Target Vessel Revascularization (TVR): number analyzed (Participants) | 277 | 98 | 52 | 12
  1-Month All Target Vessel Revascularization (TVR) | 0 | 0 | 1 | 0
  1-Month All Target Limb Amputation: number analyzed (Participants) | 277 | 98 | 52 | 12
  1-Month All Target Limb Amputation | 0 | 0 | 0 | 0
  6-Month All Deaths: number analyzed (Participants) | 275 | 96 | 52 | 12
  6-Month All Deaths | 3 | 2 | 2 | 1
  6-Month All Target Lesion Revascularization (TLR): number analyzed (Participants) | 275 | 96 | 52 | 12
  6-Month All Target Lesion Revascularization (TLR) | 2 | 3 | 1 | 0
  6-Month All Target Vessel Revascularization (TVR): number analyzed (Participants) | 275 | 96 | 52 | 12
  6-Month All Target Vessel Revascularization (TVR) | 3 | 3 | 1 | 0
  6-Month All Target Limb Amputation: number analyzed (Participants) | 275 | 96 | 52 | 12
  6-Month All Target Limb Amputation | 1 | 0 | 0 | 0
  12- Month All Deaths: number analyzed (Participants) | 259 | 93 | 52 | 12
  12- Month All Deaths | 5 | 2 | 3 | 1
  12-Month All Target Lesion Revascularization (TLR): number analyzed (Participants) | 259 | 93 | 52 | 12
  12-Month All Target Lesion Revascularization (TLR) | 14 | 15 | 3 | 2
  12-Month All Target Vessel Revascularization (TVR): number analyzed (Participants) | 259 | 93 | 52 | 12
  12-Month All Target Vessel Revascularization (TVR) | 16 | 15 | 3 | 3
  12-Month All Target Limb Amputation: number analyzed (Participants) | 259 | 93 | 52 | 12
  12-Month All Target Limb Amputation | 1 | 0 | 0 | 1
  24-Month All Deaths: number analyzed (Participants) | 254 | 90 | 0 | 12
  24-Month All Deaths | 14 | 3 |  | 1
  24-Month All Target Lesion Revascularization (TLR): number analyzed (Participants) | 254 | 90 | 0 | 12
  24-Month All Target Lesion Revascularization (TLR) | 32 | 19 |  | 3
  24-Month All Target Vessel Revascularization (TVR): number analyzed (Participants) | 254 | 90 | 0 | 12
  24-Month All Target Vessel Revascularization (TVR) | 38 | 20 |  | 4
  24-Month All Target Limb Amputation: number analyzed (Participants) | 254 | 90 | 0 | 12
  24-Month All Target Limb Amputation | 1 | 1 |  | 1
  36-Month All Deaths: number analyzed (Participants) | 249 | 88 | 0 | 11
  36-Month All Deaths | 29 | 5 |  | 1
  36-Month All Target Lesion Revascularization (TLR): number analyzed (Participants) | 249 | 88 | 0 | 11
  36-Month All Target Lesion Revascularization (TLR) | 42 | 21 |  | 3
  36-Month All Target Vessel Revascularization (TVR): number analyzed (Participants) | 249 | 88 | 0 | 11
  36-Month All Target Vessel Revascularization (TVR) | 49 | 23 |  | 4
  36-Month All Target Limb Amputation: number analyzed (Participants) | 249 | 88 | 0 | 11
  36-Month All Target Limb Amputation | 1 | 3 |  | 1
  48-Month All Deaths: number analyzed (Participants) | 242 | 84 | 0 | 10
  48-Month All Deaths | 36 | 10 |  | 2
  48-Month All Target Lesion Revascularization (TLR): number analyzed (Participants) | 242 | 84 | 0 | 10
  48-Month All Target Lesion Revascularization (TLR) | 52 | 23 |  | 3
  48-Month All Target Vessel Revascularization (TVR): number analyzed (Participants) | 242 | 84 | 0 | 10
  48-Month All Target Vessel Revascularization (TVR) | 60 | 26 |  | 4
  48-Month All Target Limb Amputation: number analyzed (Participants) | 242 | 84 | 0 | 10
  48-Month All Target Limb Amputation | 2 | 3 |  | 1
  60-Month All Deaths: number analyzed (Participants) | 248 | 85 | 0 | 10
  60-Month All Deaths | 40 | 16 |  | 2
  60-Month All Target Lesion Revascularization (TLR): number analyzed (Participants) | 248 | 85 | 0 | 10
  60-Month All Target Lesion Revascularization (TLR) | 56 | 23 |  | 3
  60-Month All Target Vessel Revascularization (TVR): number analyzed (Participants) | 248 | 85 | 0 | 10
  60-Month All Target Vessel Revascularization (TVR) | 64 | 26 |  | 4
  60-Month All Target Limb Amputation: number analyzed (Participants) | 248 | 85 | 0 | 10
  60-Month All Target Limb Amputation | 3 | 3 |  | 1

8. Secondary Outcome: Number of Participants With Rate of Primary Sustained Clinical Improvement as Assessed by Changes in Rutherford Classification From Baseline
Description: Endpoint determined to be a success when there is an improvement in Rutherford Classification of one or more categories as compared to pre-procedure without the need for repeat TLR.
  LB Substudy: Follow-up through 12-month. PK Substudy: There was no prespecified analysis of Rate of Primary Sustained Clinical Improvement for PK substudy.
Time Frame: 1, 6, 12, 24 and 36 months post-procedure (RCT); 1, 6 and 12 months post-procedure (LB substudy).
Population: Primary sustained clinical improvement rates are based on number of evaluable subjects - subjects with the data point collected.
  LB Substudy: Follow-up through 12-month. PK Substudy: There was no prespecified analysis of Rate of Primary Sustained Clinical Improvement for PK substudy.
Measure: Count of Participants; unit: Participants
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT | Long Balloon (LB) Substudy
Number analyzed (Participants) | 278 | 98 | 52
Participants
  1-Month Primary Sustained Clinical Improvement: number analyzed (Participants) | 272 | 97 | 52
  1-Month Primary Sustained Clinical Improvement | 256 | 91 | 50
  6-Month Primary Sustained Clinical Improvement: number analyzed (Participants) | 263 | 91 | 49
  6-Month Primary Sustained Clinical Improvement | 249 | 83 | 48
  12-Month Primary Sustained Clinical Improvement: number analyzed (Participants) | 252 | 91 | 48
  12-Month Primary Sustained Clinical Improvement | 222 | 69 | 45
  24-Month Primary Sustained Clinical Improvement: number analyzed (Participants) | 224 | 83 | 0
  24-Month Primary Sustained Clinical Improvement | 180 | 59 |
  36-Month Primary Sustained Clinical Improvement: number analyzed (Participants) | 198 | 72 | 0
  36-Month Primary Sustained Clinical Improvement | 150 | 53 |

9. Secondary Outcome: Number of Participants With Rate of Secondary Sustained Clinical Improvement as Assessed by Changes in Rutherford Classification From Baseline.
Description: Endpoint determined to be a success when there is an improvement in Rutherford Classification of one or more categories as compared to pre-procedure including those subjects with repeat TLR.
  LB Substudy: Follow-up through 12-months. PK Substudy: There was no prespecified analysis of Rate of Secondary Sustained Clinical Improvement for PK substudy.
Time Frame: 1, 6, 12, 24 and 36 months post-procedure (RCT): 1, 6, and 12 months post-procedure (LB substudy)
Population: Secondary sustained clinical improvement rates are based on number of evaluable subjects - subjects with the data point collected.
  LB Substudy: Follow-up through 12-months. PK Substudy: There was no prespecified analysis of Rate of Secondary Sustained Clinical Improvement for PK substudy.
Measure: Count of Participants; unit: Participants
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT | Long Balloon (LB) Substudy
Number analyzed (Participants) | 278 | 98 | 52
Participants
  1-Month Secondary Sustained Clinical Improvement: number analyzed (Participants) | 272 | 97 | 52
  1-Month Secondary Sustained Clinical Improvement | 256 | 91 | 51
  6-Month Secondary Sustained Clinical Improvement: number analyzed (Participants) | 263 | 91 | 49
  6-Month Secondary Sustained Clinical Improvement | 251 | 85 | 48
  12-Month Secondary Sustained Clinical Improvement: number analyzed (Participants) | 252 | 91 | 48
  12-Month Secondary Sustained Clinical Improvement | 230 | 81 | 47
  24-Month Secondary Sustained Clinical Improvement: number analyzed (Participants) | 224 | 83 | 0
  24-Month Secondary Sustained Clinical Improvement | 205 | 73 |
  36-Month Secondary Sustained Clinical Improvement: number analyzed (Participants) | 198 | 72 | 0
  36-Month Secondary Sustained Clinical Improvement | 176 | 67 |

10. Secondary Outcome: Number of Participants With Rate of Hemodynamic Improvement as Assessed by Changes in Ankle Brachial Index (ABI) From Baseline.
Description: Improvement of ABI by ≥ 0.1 or to an ABI ≥ 0.90 as compared to the pre-procedure value without the need for repeat revascularization.
  LB Substudy: Follow-up through 12-months. PK Substudy: There was no prespecified analysis of Rate of Hemodynamic Improvement for PK substudy.
Time Frame: 1, 6, 12, 24, and 36 months post-procedure (RCT); 1, 6, and 12 months post-procedure (LB substudy)
Population: Hemodynamic improvement rates are based on number of evaluable subjects - subjects with the data point collected.
  LB Substudy: Follow-up through 12-months. PK Substudy: There was no prespecified analysis of Rate of Hemodynamic Improvement for PK substudy.
Measure: Count of Participants; unit: Participants
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT | Long Balloon (LB) Substudy
Number analyzed (Participants) | 278 | 98 | 52
Participants
  1-Month Hemodynamic Improvement: number analyzed (Participants) | 271 | 92 | 46
  1-Month Hemodynamic Improvement | 252 | 83 | 43
  6-Month Hemodynamic Improvement: number analyzed (Participants) | 259 | 87 | 45
  6-Month Hemodynamic Improvement | 230 | 66 | 43
  12-Month Hemodynamic Improvement: number analyzed (Participants) | 251 | 84 | 43
  12-Month Hemodynamic Improvement | 202 | 57 | 40
  24-Month Hemodynamic Improvement: number analyzed (Participants) | 220 | 78 | 0
  24-Month Hemodynamic Improvement | 166 | 47 |
  36-Month Hemodynamic Improvement: number analyzed (Participants) | 196 | 69 | 0
  36-Month Hemodynamic Improvement | 128 | 45 |

11. Secondary Outcome: Walking Improvement (Distance) at 6 and 12 Months as Assessed by Change in Six Minute Walk Test (6MWT) From Baseline
Description: The 6MWT measure the maximal walking distance that a patient achieves on a flat, hard surface within a period of 6 minutes. It evaluates the global and integrated responses of all physiological systems involved during exercise including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, neuromuscular units and muscle metabolism. Change in distance walked from baseline to 12 months.
  LB Substudy: There was no prespecified analysis of Walking Improvement (distance) for the LB substudy.
  PK Substudy: There was no prespecified analysis of Walking Improvement (distance) for PK substudy.
Time Frame: 6 and 12 months post-procedure (RCT)
Population: Data provided is total distance walked (m) change from baseline. Walking Improvement (distance) assessed by change in Six Minute Walk Test (6MWT) is based on number of evaluable subjects - subjects with data point collected.
  LB Substudy: There was no prespecified analysis of Walking Improvement (distance) for the LB substudy.
  PK Substudy: There was no prespecified analysis of Walking Improvement (distance) for PK substudy.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT
Number analyzed (Participants) | 278 | 98
Meters
  6-Month Walking Improvement (Distance): number analyzed (Participants) | 252 | 84
  6-Month Walking Improvement (Distance) | 40.7 (179.0) | 55.9 (117.5)
  12-Month Walking Improvement (Distance): number analyzed (Participants) | 235 | 88
  12-Month Walking Improvement (Distance) | 36.3 (162.2) | 46.1 (115.4)

12. Secondary Outcome: Walking Improvement Assessed by Change in Walking Impairment Questionnaire (WIQ) From Baseline.
Description: The WIQ is a functional assessment questionnaire that evaluates walking ability with regard to speed, distance and stair climbing ability. It also assesses the reasons that walking ability might be limited. Range of scores include 0% (worst score) to 100% (best score). Walking improvement change assessed from baseline.
  LB Substudy: There was no prespecified analysis of Walking Improvement for the LB substudy.
  PK Substudy: There was no prespecified analysis of Walking Improvement for the PK substudy.
Time Frame: 1, 6, 12, 24 and 36 months post-procedure (RCT)
Population: Walking improvement rates are based on number of evaluable subjects - subjects with the data point collected.
  LB Substudy: There was no prespecified analysis of Walking Improvement for the LB substudy.
  PK Substudy: There was no prespecified analysis of Walking Improvement for the PK substudy.
Measure: Mean (Standard Deviation); unit: Percentage increase
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT
Number analyzed (Participants) | 278 | 98
Percentage increase
  1-Month Walking Improvement Scoring Summary: number analyzed (Participants) | 270 | 95
  1-Month Walking Improvement Scoring Summary | 33.61 (35.78) | 34.47 (35.20)
  6-Month Walking Improvement Scoring Summary: number analyzed (Participants) | 262 | 89
  6-Month Walking Improvement Scoring Summary | 32.25 (37.07) | 32.25 (37.07)
  12-Month Walking Improvement Scoring Summary: number analyzed (Participants) | 248 | 90
  12-Month Walking Improvement Scoring Summary | 32.06 (39.49) | 34.72 (36.85)
  24-Month Walking Improvement Scoring Summary: number analyzed (Participants) | 222 | 84
  24-Month Walking Improvement Scoring Summary | 29.50 (36.87) | 29.76 (41.88)
  36-Month Walking Improvement: number analyzed (Participants) | 205 | 73
  36-Month Walking Improvement | 30.37 (38.85) | 34.93 (39.03)

13. Secondary Outcome: Duplex-defined Binary Restenosis (PSVR > 2.4) of the Target Lesion
Description: Duplex-defined binary restenosis (PSVR > 2.4) of the target lesion at 1, 6, 12, 24 and 36 Months (RCT) Duplex-defined binary restenosis (PSVR > 2.4) of the target lesion at 1, 6, and 12 (LB Substudy)
  PK Substudy: There was no prespecified analysis of duplex defined binary restenosis of the target lesion
Time Frame: 1, 6, 12, 24, and 36-months post-procedure (RCT); 1, 6, and 12-months post-procedure (LB substudy)
Population: Only subjects with Diagnostic and readable PSVR values are included in the analysis.
  PK Substudy: There was no prespecified analysis of duplex defined binary restenosis of the target lesion
Measure: Count of Participants; unit: Participants
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT | Long Balloon (LB) Substudy
Number analyzed (Participants) | 278 | 98 | 52
Participants
  1-month PSVR > 2.4: number analyzed (Participants) | 179 | 63 | 38
  1-month PSVR > 2.4 | 7 | 0 | 3
  6-month PSVR > 2.4: number analyzed (Participants) | 175 | 58 | 40
  6-month PSVR > 2.4 | 8 | 12 | 2
  12-month PSVR > 2.4: number analyzed (Participants) | 177 | 59 | 41
  12-month PSVR > 2.4 | 21 | 8 | 3
  24-month PSVR > 2.4: number analyzed (Participants) | 160 | 60 | 0
  24-month PSVR > 2.4 | 17 | 6 |
  36-month PSVR > 2.4: number analyzed (Participants) | 130 | 48 | 0
  36-month PSVR > 2.4 | 17 | 5 |

14. Secondary Outcome: Patient Utility Values as Assessed by Change in EQ-5D From Baseline.
Description: Patient Utility Values as assessed by change in EQ-5D from baseline at 1, 6, 12, 24 and 36-months post-procedure. The EuroQOL (EQ)-5D is a multi-attribute health classification system. The EQ-5D uses a 5-dimension (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) descriptive system, which each consisting of 5 response options (no problems, slight problems, moderate problems, severe problems, or extreme problems/inability to perform). Outcomes reported as "Improvement" defined as improving at least one category from baseline.
  LB Substudy: There was no prespecified analysis of Patient Utility Values for the LB Substudy.
  PK Substudy: There was no prespecified analysis of Patient Utility Values for the PK Substudy.
Time Frame: 1, 6, 12, 24 and 36-months post-procedure (RCT).
Population: Patient Utility Value improvement rates are based on number of evaluable subjects - subjects with the data point collected.
  LB Substudy: There was no prespecified analysis of Patient Utility Values for the LB Substudy.
  PK Substudy: There was no prespecified analysis of Patient Utility Values for the PK Substudy.
Measure: Count of Participants; unit: Participants
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT
Number analyzed (Participants) | 278 | 98
Participants
  1-Month Mobility Improvement: number analyzed (Participants) | 270 | 95
  1-Month Mobility Improvement | 149 | 52
  1-Month Self-Care Improvement: number analyzed (Participants) | 270 | 95
  1-Month Self-Care Improvement | 24 | 12
  1-Month Usual Activities Improvement: number analyzed (Participants) | 270 | 95
  1-Month Usual Activities Improvement | 107 | 44
  1-Month Pain/Discomfort Improvement: number analyzed (Participants) | 270 | 95
  1-Month Pain/Discomfort Improvement | 141 | 61
  1-Month Anxiety/Depression Improvement: number analyzed (Participants) | 270 | 95
  1-Month Anxiety/Depression Improvement | 55 | 23
  6-Months Mobility Improvement: number analyzed (Participants) | 262 | 89
  6-Months Mobility Improvement | 149 | 45
  6-Month Self-Care Improvement: number analyzed (Participants) | 262 | 89
  6-Month Self-Care Improvement | 27 | 10
  6-Month Usual Activities Improvement: number analyzed (Participants) | 262 | 89
  6-Month Usual Activities Improvement | 102 | 38
  6-Month Pain/Discomfort Improvement: number analyzed (Participants) | 262 | 89
  6-Month Pain/Discomfort Improvement | 126 | 47
  6-Month Anxiety/Depression Improvement: number analyzed (Participants) | 262 | 89
  6-Month Anxiety/Depression Improvement | 61 | 24
  12-Months Mobility Improvement: number analyzed (Participants) | 248 | 90
  12-Months Mobility Improvement | 140 | 48
  12-Month Self-Care Improvement: number analyzed (Participants) | 248 | 90
  12-Month Self-Care Improvement | 26 | 14
  12-Month Usual Activities Improvement: number analyzed (Participants) | 248 | 90
  12-Month Usual Activities Improvement | 94 | 41
  12-Month Pain/Discomfort Improvement: number analyzed (Participants) | 248 | 90
  12-Month Pain/Discomfort Improvement | 132 | 51
  12-Month Anxiety/Depression Improvement: number analyzed (Participants) | 248 | 90
  12-Month Anxiety/Depression Improvement | 59 | 22
  24-Months Mobility Improvement: number analyzed (Participants) | 222 | 84
  24-Months Mobility Improvement | 109 | 42
  24-Month Self-Care Improvement: number analyzed (Participants) | 222 | 84
  24-Month Self-Care Improvement | 17 | 12
  24-Month Usual Activities Improvement: number analyzed (Participants) | 222 | 84
  24-Month Usual Activities Improvement | 87 | 38
  24-Month Pain/Discomfort Improvement: number analyzed (Participants) | 222 | 84
  24-Month Pain/Discomfort Improvement | 108 | 48
  24-Month Anxiety/Depression Improvement: number analyzed (Participants) | 222 | 84
  24-Month Anxiety/Depression Improvement | 47 | 17
  36-Months Mobility Improvement: number analyzed (Participants) | 206 | 73
  36-Months Mobility Improvement | 100 | 37
  36-Month Self-Care Improvement: number analyzed (Participants) | 206 | 73
  36-Month Self-Care Improvement | 17 | 8
  36-Month Usual Activities Improvement: number analyzed (Participants) | 206 | 73
  36-Month Usual Activities Improvement | 80 | 32
  36-Month Pain/Discomfort Improvement: number analyzed (Participants) | 206 | 73
  36-Month Pain/Discomfort Improvement | 96 | 38
  36-Month Anxiety/Depression Improvement: number analyzed (Participants) | 206 | 73
  36-Month Anxiety/Depression Improvement | 54 | 16

15. Secondary Outcome: Changes in Healthcare Utilization Over Time
Description: Changes in healthcare utilization over time as measured by hospitalization readmission.
  Readmission Rate represents (# of subjects/Total enrolled subjects) who were hospitalized due to TLR/TVR or due to Procedure/Device related AE.
  LB Substudy: Follow-up through 12 Month. PK Substudy: There was no prespecified analysis of healthcare utilization over time for the PK Substudy.
Time Frame: 1, 6, 12, 24, 36, 48 and 60-months post-procedure (RCT); 1, 6, 12-months post-procedure (LB substudy)
Population: Hospitalization readmission rates are based on number of enrolled subjects.
  LB Substudy: Follow-up through 12 Month. PK Substudy: There was no prespecified analysis of healthcare utilization over time for the PK Substudy.
Measure: Count of Participants; unit: Participants
Arm/Group | RANGER™ Paclitaxel Coated Balloon RCT | Standard Balloon Angioplasty RCT | Long Balloon (LB) Substudy
Number analyzed (Participants) | 278 | 98 | 52
Participants
  1-Month Readmission Rate | 6 | 4 | 1
  6-month Readmission Rate | 8 | 5 | 1
  12-Month Readmission Rate | 18 | 9 | 3
  24-Month Readmission Rate: number analyzed (Participants) | 278 | 98 | 0
  24-Month Readmission Rate | 28 | 13 |
  36-month Readmission Rate: number analyzed (Participants) | 278 | 98 | 0
  36-month Readmission Rate | 33 | 15 |
  48-Month Readmission Rate: number analyzed (Participants) | 278 | 98 | 0
  48-Month Readmission Rate | 37 | 16 |
  60-Month Readmission Rate: number analyzed (Participants) | 278 | 98 | 0
  60-Month Readmission Rate | 41 | 16 |

16. Secondary Outcome: PK Parameters Paclitaxel (PTx) Dose
Description: Summary of Pharmacokinetic Parameters in PK substudy. Paclitaxel (PTx) Dose
  PK parameter data not collected or analyzed in RCT or LB substudy.
Time Frame: Time points for analysis are a venous blood draw at screening, followed by blood draws at 10 minutes, 30 minutes, 1 hour, 3 hours, 6 hours and 24 or 48 hours after last Ranger DCB balloon removal, as well as 7 days and 30 days post index procedure.
Population: PK parameter data not collected or analyzed in RCT or LB substudy.
Measure: Mean (Standard Deviation); unit: μg
Arm/Group | Pharmacokinetics (PK) Substudy
Number analyzed (Participants) | 12
μg | 6136.6 (2554.3)

17. Secondary Outcome: PK Parameters - Maximum Plasma Concentration
Description: Summary of Pharmacokinetic Parameters in PK substudy. cmax (ng/mL) = Maximum plasma concentration
  PK data not collected or analyzed in RCT or LB substudy.
Time Frame: as for outcome 16
Population: PK data not collected or analyzed in RCT or LB substudy.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pharmacokinetics (PK) Substudy
Number analyzed (Participants) | 12
ng/mL | 2.50 (2.17)

18. Secondary Outcome: PK Parameters - Tmax
Description: Summary of Pharmacokinetic Parameters in PK substudy. - Tmax Tmax (h) = The timepoint where cmax is reached
  PK parameter data not collected or analyzed in RCT or LB substudy.
Time Frame: as for outcome 16
Population: PK data not collected or analyzed in RCT or LB substudy.
Measure: Mean (Standard Deviation); unit: hours (h)
Arm/Group | Pharmacokinetics (PK) Substudy
Number analyzed (Participants) | 12
hours (h) | 0.17 (0)

19. Secondary Outcome: PK Parameters - Area Under the Blood Concentration Versus Time Curve From Time Zero up to the Time of the Last Quantifiable Concentration, Calculated by Trapezoidal Methods.
Description: Summary of Pharmacokinetic Parameters in PK substudy. AUC0-t (ng*h/mL) = Area under the blood concentration versus time curve from time zero up to the time of the last quantifiable concentration, calculated by trapezoidal methods.
  PK parameter data not collected or analyzed in RCT or LB substudy.
Time Frame: as for outcome 16
Population: PK data not collected or analyzed in RCT or LB substudy.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Pharmacokinetics (PK) Substudy
Number analyzed (Participants) | 12
ng*h/mL | 0.86 (0.76)

ADVERSE EVENTS:
Time Frame: Adverse event data collected through five-year (60-month) post-index procedure in RCT and PK substudy. Adverse event data collected through 12-month post index procedure in LB substudy All-Cause crude mortality includes deaths confirmed through survival status assessments.
Description: RCT: 5 year data displayed PK Substudy: 5 year data displayed; PK substudy: Adverse events are collected as required in RCT but not analyzed.
  LB Substudy: 12 month data displayed
Groups:
- RANGER™ Paclitaxel Coated Balloon: RANGER™ Paclitaxel Coated Balloon Catheter angioplasty in the SFA/PPA at the index procedure.
- Standard Balloon Angioplasty: Standard Balloon Catheter angioplasty in the SFA/PPA at the index procedure.
Arm/Group | RANGER™ Paclitaxel Coated Balloon | Standard Balloon Angioplasty | Long Balloon (LB) Substudy | Pharmacokinetics (PK) Substudy
All-Cause Mortality (participants affected / at risk) | 44/278 | 20/98 | 2/52 | 3/12
Serious Adverse Events (participants affected / at risk) | 212/278 | 73/98 | 23/52 | 10/12
Other Adverse Events (participants affected / at risk) | 176/278 | 63/98 | 26/52 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RANGER™ Paclitaxel Coated Balloon (N=278) | Standard Balloon Angioplasty (N=98) | Long Balloon (LB) Substudy (N=52) | Pharmacokinetics (PK) Substudy (N=12)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 1 (1) | 0 (0) | 3 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 7 (8) | 7 (7) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 11 (11) | 3 (3) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 8 (8) | 2 (2) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 9 (14) | 2 (3) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 10 (16) | 4 (4) | 1 (1) | 1 (3)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 9 (11) | 4 (8) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 12 (13) | 4 (6) | 1 (2) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 4 (5) | 3 (4) | 2 (3) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
Eyelid cyst (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 (9) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 5 (5) | 1 (1) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Accidental death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Device related thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Implant site inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (2)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 4 (6) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 15 (18) | 9 (9) | 4 (4) | 3 (6)
Post procedural infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 4 (5) | 3 (3) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 2 (2) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery bypass graft stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 4 (4) | 1 (2) | 0 (0) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 11 (11) | 5 (5) | 2 (2) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 0 (0) | 1 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Mylagia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (3) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Plantar fascitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 6 (7) | 2 (2) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (4) | 3 (3) | 0 (0) | 0 (0)
Dementia with Lewy bodies (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 11 (16) | 4 (6) | 0 (0) | 2 (2)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 6 (9) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (7) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Angiodysplasia (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 32 (48) | 9 (11) | 0 (0) | 1 (1)
Lower limb artery perforation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 14 (24) | 8 (13) | 0 (0) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 22 (31) | 9 (11) | 1 (1) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 63 (109) | 18 (38) | 7 (9) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 11 (16) | 2 (2) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Hyperstensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular stent stenosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular stent occlusion (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Coronary artery perforation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac sarcoidosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 5 (5) | 1 (2) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric mucosal lesion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 1 (3) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chemical peritonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethral haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 3 (4) | 3 (4) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Cervical myelopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Investigations) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Splenic haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Macular fibrosis (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cataract nuclear (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ectropion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Organic erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RANGER™ Paclitaxel Coated Balloon (N=278) | Standard Balloon Angioplasty (N=98) | Long Balloon (LB) Substudy (N=52) | Pharmacokinetics (PK) Substudy (N=12)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thyroglossal cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocrine ophthalmopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heterophoria (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mydriasis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pterygium (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melanosis coli (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 6 (6) | 2 (3) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 7 (7) | 3 (3) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tenderness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 5 (6) | 2 (2) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulval abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 0 (0) | 1 (1)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 11 (11) | 2 (2) | 1 (1) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Ankle brachial index decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid bruit (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lipids abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulse absent (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Right ventricular systolic pressure (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ultrasound Doppler abnormal (Investigations) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 4 (4) | 2 (2) | 4 (4)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (16) | 7 (7) | 2 (2) | 0 (0)
Plantar fascitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular carinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 5 (6) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postural tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Middle insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (6) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epiglottic mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic pigmented purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blue toe syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 9 (10) | 3 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 31 (37) | 11 (13) | 2 (2) | 1 (1)
Internal haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 17 (18) | 6 (6) | 6 (6) | 2 (2)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subclavian steal syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic limb pain (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT03064126/Prot_SAP_000.pdf